CLINICAL TRIAL: NCT06908018
Title: Safety, Virological and Immunological Assessment of the Controlled Dengue Human Infection Model in Dengue-Immune Participants in Thailand (DHIT-Immune)
Acronym: DHIT-Immune
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MU-MOU780/2567(IRB1)
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Safety Issues; Dengue; Viremia; Immune-related Adverse Event
MeSH Terms: conditions — Dengue; Viremia

STUDY DESIGN:
Intervention Model Description: Challenge the attenuated virus in 12 dengue-immune participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label DENV2delta30 virus challenge (Experimental)
  Interventions: Biological: rDEN2Δ30-7169

INTERVENTIONS:
Biological: rDEN2Δ30-7169 — rDEN2Δ30-7169 is a recombinat virus that could induce viremia and immunological responses with out serious adverse effect. The virus will be challenged after participants screening and consent for hospitalization. After virus challenge, the virological, immunological and clinical manifestation will be recorded and analyzed for the result from day 0-60 post-virus challenge.

SUMMARY:
rDEN2Δ30-7169 is a dengue challenge strain that previously reports its viremia induction effect in participants with minimal symptoms in US flavivirus naïve participants. Moreover, preliminary result of five Thai dengue naïve participants from previous project (registered number NCT05476757) demonstrated 100% viremia status without severe adverse event after 60 days post-virus challenge. However, result from previous project may not fully represent the clinical manifestation and immunological responses of major population of endemic areas, where most people in endemic area have dengue immune status. Therefore, this controlled human infection model protocol proposes to challenge the attenuated virus in 12 dengue-immune participants recruited from Bangkok metropolitan area, Thailand. We aim to assess the safety, viremia, NS1 antigenemia profile, and immunogenicity of the challenge virus in the dengue immune participants. After finish safety assessment, all participants will be vaccinated with a full course of dengue vaccines to prevent recurrent dengue infection. Immunological responses after vaccination will be also evaluated the vaccine efficacy.

Our expected outcomes are all participants present viremia profiles after virus challenge without serious adverse events (SAE). The exploratory profiles include assesment of immune profiles and parameters comparison with the other dengue challenge study.

ELIGIBILITY:
Inclusion Criteria:

1. Thai healthy volunteers, aged between 18 to 40 years old, weight is greater than or equal to 50 kg and have Thai language literacy.
2. Have not given blood donation in the past 3 months.
3. Education: high school diploma or above
4. Positive dengue-immune status against DENV-1 and/or DENV-3 and/or DENV-4 with naive DENV-2 status by the standard FRNT 50% (FRNT50) as follows: FRNT50 titer against

   * DENV1 ≥ 1:5 and/or
   * DENV3 ≥ 1:5 and/or
   * DENV4 ≥ 1:5 with
   * DENV2 ≤ 1:16
5. Willingness to participate in the study as evidenced by signing the informed consent document.
6. Female participants of childbearing potential should be agreed to either abstinence or use at least one primary form of contraception from the time of screening for rDEN2Δ30-7169 administration until 1 month after complete course of Dengue vaccination (Study Day 298).

Exclusion Criteria:

1. For female participants: Currently pregnant, as determined by positive urine human choriogonadotropin (HCG) test or breast-feeding, and given birth or abortion within 6 months.
2. History of previous acute undifferentiated febrile illness leading to hospitalization in the past 3 months.
3. Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the requirements of the study protocol.
4. Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
5. History of a severe allergic reaction or anaphylaxis.
6. Severe asthma (emergency room visit or hospitalization within the last 6 months).
7. Any known immunodeficiency syndrome.
8. Having any pre-existing medical conditions consist of thrombocytopenia, autoimmune disease and cancer based on history, physical examination, and/or laboratory studies.
9. Current use of anticoagulant medications (this includes anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
10. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. An immunosuppressive dose of corticosteroids is defined as ≥ 10 mg of a prednisone equivalent per day for ≥ 14 days.
11. Asplenia
12. Receipt of any vaccine within 28 days or a killed vaccine within 14 days prior to receiving virus administration, or anticipated receipt of any vaccine during the 28 days following rDEN2Δ30-7169 administration.
13. Has an obvious history of receiving any type of dengue vaccine or has previously participated in dengue vaccine research.
14. Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following rDEN2Δ30-7169 administration.
15. History of allergy to Qdenga vaccine or any components of the vaccine.
16. Previous episode of severe dengue infection defined by WHO 2009
17. Screening laboratory values of Grade 1 or above (as defined in this protocol) for ANC (<750 /mm3), Platelet (<100,000 /mm3), PT (> 1.25 x ULN), APTT (> 1.66 x ULN), ALT (>2.5 x ULN) and plasma creatinine (> 1.3 x ULN OR Increase to >1.3 x participant's baseline).
18. A participant with hemoglobin level less than 10 g/dL at initial screening.
19. Body temperature is greater than or equal to 38.0 °C (Oral)
20. HIV infection, as indicated by anti-HIV screening assays.
21. Hepatitis C virus (HCV) infection, as indicated by anti-HCV screening assays.
22. Hepatitis B virus (HBV) infection, as indicated by hepatitis B surface antigen (HBsAg) and/or anti-HBc screening.
23. Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The safety of rDEN2Δ30-7169 in Dengue immune participants | Day 0 -60 after virus challenge
  To evaluate the safety of rDEN2Δ30-7169 in dengue-immune participants as assessed by the frequency of virus-related adverse events (AEs), graded by severity.

IPD SHARING:
Plan to Share IPD: No